CLINICAL TRIAL: NCT00405145
Title: Mapping of the Eloquent Cortex and of Epileptic Networks Using Functional Magnetic Resonance Imaging and Electroencephalography in Epileptic Patients
Brief Title: Mapping of the Epileptic Brain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Other Study IDs: 0618
Record Dates: First submitted 2006-08-07; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; MRI; EEG; Neuroimaging
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study aims improving the outcome after brain resective surgery of epileptic patients by improving presurgical evaluations. In particular the specific goal is to evaluate the ability of non invasive neuroimaging (functional magnetic resonance imaging and electroencephalography) to provide presurgical maps of the functional areas of the brain and of the epileptogenic networks.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy

Exclusion Criteria:

* MRI incompatible
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-07; Study Completion 2011-07

CONTACTS AND LOCATIONS:
Overall Officials: Olivier David, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Jean-François Le Bas, MD, PhD, Principal Investigator — University Grenoble Hospital
Locations (1):
- UniversityHospitalGrenoble, Grenoble, ISERE, France